CLINICAL TRIAL: NCT01267539
Title: Suan Tsao Jen Tang for Treating Menopause With Sleep Problem: a Clinical Observation
Status: Completed | Type: Observational
Sponsor: Taipei City Hospital (Other Government)
Collaborators: Chinese Medical Association (Network)
Responsible Party: Jung-Lien Lai/Taipei City Hospital, Taipei City Hospital
Other Study IDs: TCHIRB-970110-E
Record Dates: First submitted 2010-12-20; First posted 2010-12-28 (Estimated); Last update posted 2010-12-28 (Estimated); Status verified 2008-01

CONDITIONS: Menopausal and Female Climacteric States
Keywords: Suan Zao Ren Tang, climacteric, PSQI, WHOQOL-BREF

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
A prospective follow-up study was carried out in the Yang Ming branch of the Taipei City Hospital.Climacteric women with sleep difficulty received SZRT at a rate of 4.0 g, thrice daily for four weeks.

DETAILED DESCRIPTION:
A prospective follow-up study was carried out in the Yang Ming branch of the Taipei City Hospital between April 2008 and April 2010. Sixty-seven climacteric women with sleep difficulty received SZRT at a rate of 4.0 g, thrice daily for four weeks. Baseline scores were measured on the Pittsburg Sleep Quality Index (PSQI), followed by further measures at the end of weeks one and four. The World Health Organization Quality of Life (WHOQOL) assessment and the Menopause Rating Scale (MRS) were undertaken as secondary outcomes. Regression models were constructed to explore the score differences between the baseline and at weeks one and four by various determinants including age, body mass index (BMI), and severity of baseline menopausal symptoms. Among 99 surveyed patients, 67 and 61 were screened for intention to treat (ITT) and per-protocol population set analysis, respectively. Statistically significant reductions in the PSQI index scores evidenced on the fourth week.

ELIGIBILITY:
Inclusion Criteria:

1. Climacteric women, ranging from 40-65 years of age
2. Pittsburg Sleep Quality Index (PSQI) of greater than six
3. Falling asleep more than 45 minutes or slept less than six hours

Exclusion Criteria:

1. Within three months of the study there had been a major incident
2. Working the nightshift
3. Lack of time or timing conflicts
4. Pychosis, severe depression, obstructive sleep apnea-hypopnea, cardiac arrhythmia, acute myocardial infarction, high blood pressure, diabetes, or cancer
5. Currently taking pharmaceuticals that affect melatonin, acetylcholine, glutamate, serotonin, norepinephrine, GABA, histamine, adenosine, or prostaglandins
6. Inability to read and fill out the forms for the study
7. Any evidence of renal or liver dysfunction as defined by a level of at least 1.5 times of the upper reference limit

Ages: 40 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: The subjects enrolled in the study were climacteric women, ranging from 40-65 years of age, with a Pittsburg Sleep Quality Index (PSQI) of greater than six. These women spent 45 minutes or more falling asleep, slept less than six hours, and had struggled with this issue continuously for at least one month.
Sampling Method: Non-Probability Sample
Enrollment: 67 (Actual)
Dates: Start 2008-04; Primary Completion 2010-04 (Actual); Study Completion 2010-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jung-Nien Lai, PHD, Study Chair — Taipei City Hospital
Locations (1):
- Taipei City Hospital, Taipei, Taiwan, Taiwan